CLINICAL TRIAL: NCT02453646
Title: Analysis of CRBSI (Catheter-Related Blood Stream Infection) Rates in Patients With a NexSite™ HD (Hemodialysis) Catheter
Brief Title: Analysis of CRBSI Rates in Patients With a NexSite™ HD (Hemodialysis) Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marvao Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TR 0147
Record Dates: First submitted 2015-05-18; First posted 2015-05-25 (Estimated); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NexSite HD Patients (Experimental): NexSite HD patient catheter device placement
  Interventions: Device: NexSite HD Patients

INTERVENTIONS:
Device: NexSite HD Patients — Measurement of CRBSI rate and other device related adverse events in patients with NexSite HD Catheter.

SUMMARY:
A U.S. multi-centre post approval registry to analyse the CRBSI rate in patients with the NexSite HD Catheter for long term vascular access for hemodialysis.

DETAILED DESCRIPTION:
This is a U.S. multi - centre, prospective, non-randomized post approval registry. Approximately one hundred and twenty patients will be implanted with a NexSite HD catheter at four to eight U.S. sites where hemodialysis catheters are routinely implanted. Each site may enrol a maximum of 50 patients. Enrolled patients will be followed from device placement to device removal or 180 days post device placement. Patients will be enrolled once only.

The primary endpoint is CRBSI rate related to the NexSite HD catheter. Determination of infection will be decided by the investigator and if necessary adjudicated by the CEC (Clinical Events Committee) based on blood culture results, regardless of whether the catheter is removed.

Secondary endpoints for the study are

* Successful placement and continued use of the NexSite HD device designed for use in patients requiring long term hemodialysis.
* Healing of catheter exit site
* Tunnel Infections
* Exit site infections
* Early non-infectious complications associated with CVCs
* Late non-infectious complications associated with Central Venous Catheters

ELIGIBILITY:
Inclusion Criteria:

1. The patient shall be 18 - 80 years old.
2. The patient requires the placement of a long term tunnelled HD catheter for administration of hemodialysis.
3. The patient has anticipated survival in excess of 90 days from the anticipated date of catheter placement.
4. The patient has the ability to understand the research subject information and sign a written Informed Consent form which must be obtained prior to initiation of the study.
5. The patient receives the catheter via the internal jugular or subclavian vein.
6. All female patients of child bearing potential must complete a negative pregnancy test and will confirm that they are not breastfeeding.

Exclusion Criteria:

1. The patient is participating in another IRB (Institutional Review Board) clinical trial, which modifies standard-of-care treatment and/or involves an investigational device or drug.
2. The patient has a confirmed or suspected infection, bacteraemia or septicaemia.
3. The patient's physiology is NOT suitable for placement of the NexSite device; this will include an examination of the anatomy at the proposed catheter exit site.
4. The patient is known or suspected to have allergies to the materials used in the construction of the device.
5. The patient has previously suffered from coagulation issues or has had vascular surgery at the proposed placement site.
6. The patient has received radiation treatment at the proposed catheter placement site.
7. The patient has severe chronic obstructive lung disease.
8. The patient is pyretic within 72 hours (temperature ≥38o C or 100.4oF) prior to placement and/or has received antimicrobial drugs within two weeks prior to catheterisation.
9. The patient is female of child bearing potential not using adequate contraception. (Adequate contraception is defined as abstinence, intrauterine device [IUD], birth control pills, or spermicidal gel with diaphragm or condom)
10. The patient has another indwelling catheter.
11. The patient has non-healing diabetic foot ulcers.
12. The patient did not give informed consent.
13. The patient would be unavailable for follow-up.
14. The patient is a permanent nursing home resident.
15. The proposed access site is not the internal jugular or subclavian vein.
16. The patient is scheduled to undergo an elective surgical procedure (other than a procedure to create a graft or fistula) within the study timeframe.
17. Any other condition that the Investigator believes should exclude the patient from the study.
18. The patient does not have English or Spanish as their first language.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with Catheter-Related Blood Stream Infection (CRBSI)(bacteremia/fungemia) as an adverse event. | Participants will be followed for the duration of catheter use or to 180 days post device placement (whichever occurs first)
  Number of participants with a confirmed CRBSI for the duration of catheter use or to 180 days post device placement (whichever occurs first)

SECONDARY OUTCOMES:
Number of participants with adverse events associated with device placement and use. | Participants will be followed for the duration of catheter use or to 180 days post device placement (whichever occurs first)
  Number of participants with adverse events associated with device placement and for the duration of catheter use or to 180 days post device placement.
Number of participants with unhealed catheter exit sites | Participants will be followed for the duration of catheter use or to 180 days post device placement (whichever occurs first)
  Number of participants with unhealed exit sites for the duration of catheter use or to 180 days post device placement (whichever occurs first)
Number of participants with tunnel infection as an adverse event | Participants will be followed for the duration of catheter use or to 180 days post device placement (whichever occurs first)
  Number of participants with a tunnel infection for the duration of catheter use or to 180 days post device placement (whichever occurs first)
Number of participants with exit site infection as an adverse event | Participants will be followed for the duration of catheter use or to 180 days post device placement (whichever occurs first)
  Number of participants with a exit site infection for the duration of catheter use or to 180 days post device placement (whichever occurs first)
Number of participants with Pneumothorax, haemothorax, arrhythmia, air embolism or arterial perforation as an adverse event. | 1 day of device placement
  Number of participants with non-infectious catheter complications within one day of placement.
Number of participants with Catheter dislodgement, Catheter tip dislodgement and catheter thrombosis as an adverse event. | Participants will be followed for the duration of catheter use or to 180 days post device placement (whichever occurs first)
  Number of participants with late non infectious complications for the duration of catheter use or to 180 days post device placement (whichever occurs first).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey G Hoggard, MD, Principal Investigator — Capital Nephrology Associates
Locations (6):
- United States (6):
  - Eastern Nephrology Associates, Greenville, North Carolina
  - Eastern Nephology Associates, New Bern, North Carolina
  - Capital Nephrology Associates, Raleigh, North Carolina
  - South Carolina Nephrology and Hypertension Center Inc, Orangeburg, South Carolina
  - Lubbock Vascular Access Centre, Lubbock, Texas
  - Renal Associates, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No